CLINICAL TRIAL: NCT02575846
Title: Clinical and Biological Outcomes of Human Milk and Formula Intake After Gastroschisis Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00056976
Record Dates: First submitted 2015-10-06; First posted 2015-10-15 (Estimated); Last update posted 2024-04-12 (Actual); Status verified 2017-06

CONDITIONS: Gastroschisis
MeSH Terms: conditions — Gastroschisis

ARMS (2):
- Human Milk (Active Comparator): Neonates fed human milk
  Interventions: Dietary Supplement: Enteral Intake - Human Milk
- Formula (Placebo Comparator): Neonates fed formula
  Interventions: Dietary Supplement: Enteral Intake - Formula

INTERVENTIONS:
Dietary Supplement: Enteral Intake - Human Milk — Comparing formula and human milk
  Arms: Human Milk
Dietary Supplement: Enteral Intake - Formula — Comparing formula and human milk
  Arms: Formula

SUMMARY:
The purpose of this study is to determine which type of food results in a shorter hospital stay and better overall outcome for babies born with gastroschisis.

ELIGIBILITY:
Inclusion Criteria:

* 1) neonates born with gastroschisis
* 2) neonatologist, surgeon, and parent (or care provider) willing to have the neonate participate in the study

Exclusion Criteria:

* 1) associated anomaly or medical concern that impacts hospital length of stay (i.e. intestinal atresia, very low birth weight(<1500 grams))
* 2) known major chromosomal abnormality

Ages: 2 Hours to 48 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 4 (Actual)
Dates: Start 2015-11-26 (Actual); Primary Completion 2016-11-11 (Actual); Study Completion 2016-11-11 (Actual)

PRIMARY OUTCOMES:
Length of Hospital Stay | One month

SECONDARY OUTCOMES:
Time to Full Enteral Feeds | Three weeks
Time on Total Parenteral Nutrition | Three weeks

CONTACTS AND LOCATIONS:
Overall Officials: Obinna O Adibe, MD, MHS, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Background] Kohler JA Sr, Perkins AM, Bass WT. Human milk versus formula after gastroschisis repair: effects on time to full feeds and time to discharge. J Perinatol. 2013 Aug;33(8):627-30. doi: 10.1038/jp.2013.27. Epub 2013 Mar 21. PMID 23519369
- [Background] Sydorak RM, Nijagal A, Sbragia L, Hirose S, Tsao K, Phibbs RH, Schmitt SK, Lee H, Farmer DL, Harrison MR, Albanese CT. Gastroschisis: small hole, big cost. J Pediatr Surg. 2002 Dec;37(12):1669-72. doi: 10.1053/jpsu.2002.36689. PMID 12483626
- [Background] Mastromarino P, Capobianco D, Campagna G, Laforgia N, Drimaco P, Dileone A, Baldassarre ME. Correlation between lactoferrin and beneficial microbiota in breast milk and infant's feces. Biometals. 2014 Oct;27(5):1077-86. doi: 10.1007/s10534-014-9762-3. Epub 2014 Jun 27. PMID 24970346
- [Background] Gomez-Llorente C, Plaza-Diaz J, Aguilera M, Munoz-Quezada S, Bermudez-Brito M, Peso-Echarri P, Martinez-Silla R, Vasallo-Morillas MI, Campana-Martin L, Vives-Pinera I, Ballesta-Martinez MJ, Gil A. Three main factors define changes in fecal microbiota associated with feeding modality in infants. J Pediatr Gastroenterol Nutr. 2013 Oct;57(4):461-6. doi: 10.1097/MPG.0b013e31829d519a. PMID 23752082